CLINICAL TRIAL: NCT03491566
Title: Comparison of Two Different Exercises on Increasing Cognitive Functions and Speed of Movement in Young Adults
Brief Title: Effects of Two Different Exercises on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Physiotherapist, Lecturer, Biruni University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: Biruni University
Record Dates: First submitted 2018-03-27; First posted 2018-04-09 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic Pilates Group (Experimental): Initial assessments of participants were made and they were taught key components of the Clinical Pilates exercises. Exercises were administered for 4 weeks, 3 days/week, 40-50 minutes/session under the supervision of a physiotherapist. Groups of 9-10 people with similar physical characteristics and fitness level for session times were created. The sessions were started with level 1 exercises requiring more support and less control. Each exercise was repeated 8-10 times; as the physical level of the participants increased, exercises progressed towards level 3 exercises requiring more attention, concentration and control. Each session consisted of an average of 10 minutes warm-up, 20 to 30 minutes of matt and 10 minutes cooling of of Clinical Pilates exercises.
  Interventions: Other: Clinic Pilates Group
- Aerobic Exercise Group (Experimental): Initial assessments of participants were made before the first session. Using an elliptical bicycle or bicycle, or treadmill under the supervision of a physiotherapist, a total of 150 minutes moderate intensity (50-70% of maximal heart rate (HRmax)) aerobic exercise in accordance with the World Health Organization's guideline was applied, 3 days/week (50 mins/session) or 5 days/week (30 mins /session) for 4 weeks. The instruments to be used for the exercises were chosen according to the preference of the individual. HRmax was calculated using the "220-years". For example; at the age of 20 years, the target heart rate was determined as 100-140 beats/min for moderate physical activity in a person with HRmax 200 beats/min.
  Interventions: Other: Aerobic Exercise Group

INTERVENTIONS:
Other: Clinic Pilates Group — Clinical Pilates exercises include "Hundreds", "One Leg Stretch", "Shoulder Bridge", "One Leg Kick", Swimming ", Double Leg Stretch", "Swan Dive" Circle "," Arm Opening "," Spine Twist "," Roll Down "exercises.
  Arms: Clinic Pilates Group
Other: Aerobic Exercise Group — Aerobic exercise with using an elliptical bike, or bike or treadmill under supervision of a physiotherapist.
  Arms: Aerobic Exercise Group

SUMMARY:
The aim of this study is to investigate the effectiveness of Pilates-based exercises on cognitive functions in comparison with aerobic exercises.

Individuals in the 4-weeks study will be divided into two groups using the Graphpad website: Clinical Pilates exercise group (Group 1), aerobic exercise group (Group 2). The sample size for each group was calculated as 24 people. Considering the possibility of %10 drops, 27 individuals will be included in each group and a total of 54 cases in the study. First, the socio-demographic information of the participants will be collected with a prepared form. Individuals will be assessed by the International Physical Activity Questionnaire-Short Form, Nelson Speed of Movement Test, Verbal Fluency Test and Stroop Test at pre-study,end of the first session and end of the study (4th week). Participants in control will be given will keep an activity lo to check their physical activity levels. SPSS package programme will be used in the analysis of the data and p<0.05 will be considered significant.

DETAILED DESCRIPTION:
Modern society adapts to the sedentary lifestyle. This global trend is a major threat to public health because inactivity is the leading cause of global mortality. In addition, low physical activity is related to risk of hypertension, obesity, type II diabetes, cancer, and many other chronic diseases.

There is evidence that regular physical activity contributes to primary and secondary prevention of various chronic diseases. It is claimed that physical activity can also affect cognitive functions, reduce dementia risk in addition to health benefits. However, studies investigating the effects on cognitive functions such as attention, learning and memory are limited.

As a method of physical activity, the effects of aerobic and resistive exercises on cognitive functions were generally investigated in the research.Pilates based exercises commonly used in recent studies and its effectiveness investigated in various fields are also a physical activity method with six principles including concentration, control, centering, flowing movement, precision and breathing. Pilates-based exercises that require mentally focusing on the targeted body region, develop body-mind connection, aim to increase the quality of movement by neuromuscular methods with directing attention to the moving part of body segment, appear to be a way to positively affect cognitive functions.

The aim of this study is to investigate the effectiveness of Pilates-based exercises on cognitive functions in comparison with aerobic exercises.

Individuals in the 4-weeks study will be divided into two groups using the Graphpad website: Clinical Pilates exercise group (Group 1), aerobic exercise group (Group 2). The Power and Sample Size version 3.1.2 (PS) programme was used to calculate the sample size. Because of the lack of "minimal clinical important difference" value for the Stroop test in the literature while the sample size calculation, the standard deviation value was set to 60 (σ) (derived from a similar study), the change in the means (δ) was set as 50 in the formula (power 80%, α 0.05). The sample size for each group was calculated as 24 people. Considering the possibility of %10 drops, 27 individuals will be included in each group and a total of 54 cases in the study. Individuals will be enrolled according to the inclusion criteria.

First, the socio-demographic information of the participants will be collected with a prepared form. Individuals will be assessed by the International Physical Activity Questionnaire-Short Form, Nelson Speed of Movement Test, Verbal Fluency Test and Stroop Test at pre-study and 4th week.

SPSS statistical program will be used for statistical analysis. The Shapiro Wilk test will be performed to determine the normal distribution suitability of the data. The difference between the continuous variables in the groups will be compared with the Independent T test. Paired Simple T-Test will be used to evaluate changes in each group before and after the program. In all analyzes p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy individual between the ages of 18-25,
* No problem with reading, writing or understanding Turkish,
* According to International Physical Activity Questionnaire Short Form being physically inactive (< 600 MET (metabolic equivalent of task)/mins),
* Volunteering and sustainability to the study.

Exclusion Criteria:

* Musculoskeletal system problems that prevent exercising,
* Cardiovascular system disorders such as myocardial infarction, angina, exercise intolerance, uncontrolled hypertension, etc. that limit effort capacity,
* Neurological disorder or cognitive dysfunction such as stroke, dementia, schizophrenia, etc.,
* Pregnancy,
* Smoking,
* Achromatopsia,
* Body Mass Index (BMI) higher > 35,
* Beck Depression Scale score ≥ 17.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Cognitive Function: Selective Attention, Information Processing Speed | 1 month
  Stroop test is one of the neuropsychological tests showing frontal lobe activity. It is used for evaluating information processing speed, interference effect and selective attention. In test, there are 4 cards. On the 1st card there are the names of the colors printed in black, on the 2nd card there are the names of the colors printed in red-blue-yellow-green, on the 3rd card there are circles of 0.4 cm in diameter printed in red, blue, yellow, green, on the 4th card there are "and, over, hard, when " words printed in red-blue-yellow-green.The test's basic scores are obtained by scoring the sections separately. Total score of test is obtained by the total time from the command "Start" to the reading of the last item of the card, the number of errors and the number of correction in subject' reaction.

SECONDARY OUTCOMES:
Hemispheric Cognitive Function | 1 month
  Verbal fluency test is used for evaluating the verbal-phonemic flow and identifying the recall of the desired words in given time by determining hemispheric cognitive functions. The test has two subgroups: "Letter Fluency Test" and "Category Fluency Test".
  The total score is the number of said words while error score is calculated with considering the word errors and repetitions.
Speed of Movement | 1 month
  It is used to measure combined reaction and speed of movement of the hands and the arms. Twenty trails are done by the subjects. The score for the combined response movement is obtained from the times at the point just above the upper edge of the hand after the catch was made. The five slowest and five fastest trails are discarded and mean of the middle ten trails are recorded as the ruler's fall distance. Reaction time is derived from the formula after putting ruler's fall distance.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Principal Investigator — Istanbul University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No